CLINICAL TRIAL: NCT07285174
Title: Shanghai Lymphoma Clinical Cohort
Status: Not yet recruiting | Type: Observational
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Zhao Weili, Dean, Ruijin Hospital
Other Study IDs: Shanghai Lymphoma Cohort
Record Dates: First submitted 2025-12-03; First posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Lymphoma; Cohort
Keywords: Lymphoma; Clinical; Cohort
MeSH Terms: conditions — Lymphoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — DNA and RNA will be retained.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Shanghai Lymphoma Clinical Cohort: Shanghai Lymphoma Clinical Cohort
  Interventions: Other: No interventions need to be specified for this study

INTERVENTIONS:
Other: No interventions need to be specified for this study — No interventions need to be specified for this study

SUMMARY:
The aim of this study is to prospectively collect clinical information on patients with lymphoma, and to explore the best therapeutic strategies in the real-world population.

DETAILED DESCRIPTION:
Lymphoma is a common hematological malignancy. This study aims to prospectively collect clinical information on patients with lymphoma, including the distribution of involved sites, clinical and molecular characteristics of different lymphoma subtypes, clinical treatment protocols, and prognosis, to explore the best therapeutic strategies in the real-world population.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 16 years (including 16 years old).
2. Patients newly diagnosed with non-Hodgkin lymphoma
3. Patients who have received systematic clinical treatment.
4. Patients with measurable lesions, at least containing one effective evaluation of efficacy.

Exclusion Criteria:

1. Patients who only receive supportive treatment.
2. Patients who cannot obtain effective evaluation data of efficacy.

Min Age: 16 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Adult patients with histologically confirmed diagnosis of non-Hodgkin lymphoma.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-12-18 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | Baseline up to data cut-off (up to approximately 1 year)
  Progression-Free Survival (PFS) will be defined from the date of starting therapy and the date of disease progression, relapse or death from any cause.

SECONDARY OUTCOMES:
Overall Survival (OS) | Baseline up to data cut-off (up to approximately 1 year)
  Overall Survival (OS) will be defined from the start date of therapy to the date of death from any cause.

IPD SHARING:
Plan to Share IPD: Undecided